CLINICAL TRIAL: NCT04752163
Title: An Open-Label Phase 1/2 Multi-Arm Study of DS-1594b as a Single-Agent and in Combination With Azacitidine and Venetoclax or Mini-HCVD for the Treatment of Patients With Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (ALL)
Brief Title: DS-1594b With or Without Azacitidine, Venetoclax, or Mini-HCVD for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: supporting/funding source decided to de-prioritize and stop development of DS-1594
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0946; NCI-2021-00603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0946 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Mesna; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A and B (DS-1594b) (Experimental): Patients with MLLr or NPM1m receive DS-1594b PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: DS-1594b
- Cohort C (DS-1594b, venetoclax, azacitidine) (Experimental): Patients receive DS-1594b PO BID on days 1-28, venetoclax PO QD on days 1-28, and azacitidine IV or SC on days 1-7. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: DS-1594b; Drug: Azacitidine; Drug: Venetoclax
- Cohort D (DS-1594b, mini-HCVD) (Experimental): Patients receive DS-1594b PO BID on days 1-28. For additional information, see trial description.
  Interventions: Drug: DS-1594b; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Biological: Filgrastim; Drug: Leucovorin; Drug: Mesna; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine
- Phase I (DS-1594b) Cohort 1 (Experimental): Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  70 mg twice daily.
  Interventions: Drug: DS-1594b
- Phase I (DS-1594b) Cohort 2 (Experimental): Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  50 mg twice daily.
  Interventions: Drug: DS-1594b
- Phase I (DS-1594b) Cohort 3 (Experimental): Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  20 mg daily.
  Interventions: Drug: DS-1594b
- Phase I (DS-1594b) Cohort 4 (Experimental): Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  50 mg daily.
  Interventions: Drug: DS-1594b
- Phase I (DS-1594b) Cohort 5 (Experimental): Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  100 mg daily.
  Interventions: Drug: DS-1594b

INTERVENTIONS:
Drug: DS-1594b — Given DS-1594b PO
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
  Arms: Cohort C (DS-1594b, venetoclax, azacitidine)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Cohort D (DS-1594b, mini-HCVD)
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Leucovorin — Given IV or PO
  Other Names: Folinic acid
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Mesna — Given IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Cohort D (DS-1594b, mini-HCVD)
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
  Arms: Cohort D (DS-1594b, mini-HCVD)
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Cohort C (DS-1594b, venetoclax, azacitidine)
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine
  Arms: Cohort D (DS-1594b, mini-HCVD)

SUMMARY:
This phase I/II trial studies the effect of DS-1594b with or without azacitidine, venetoclax, or mini-HCVD in treating patients with acute myeloid leukemia or acute lymphoblastic leukemia that has come back (recurrent) or not responded to treatment (refractory). Chemotherapy drugs, such as azacitidine, venetoclax, and mini-HCVD, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. DS-1594b may inhibit specific protein bindings that cause blood cancer. Giving DS-1594b, azacitidine, and venetoclax, or mini-HCVD may work better in treating patients with acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of DS-1594b followed by a phase II study.

PHASE I: Patients receive DS-1594b orally (PO) twice daily (BID) on days 1-28 in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are assigned to 1 of 4 cohorts.

COHORT A: Patients with MLLr receive DS-1594b PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients with NPM1m receive DS-1594b PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT C: Patients receive DS-1594b PO BID on days 1-28, venetoclax PO QD on days 1-28, and azacitidine intravenously (IV) or subcutaneously (SC) on days 1-7. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT D: Patients receive DS-1594b PO BID on days 1-28. For cycles 1, 3, 5, 7, patients also receive cyclophosphamide IV over 3 hours on days 1-3, mesna IV over 24 hours on days 1-3, vincristine IV on days 1 and 11, dexamethasone PO or IV on days 1-4 and 11-14, filgrastim SC on days 1-28, methotrexate intrathecally (IT) on day 2 of cycles 1 and 3, and cytarabine IT on day 7 of cycles 1 and 3. For cycles 2, 4, 6, 8, patients also receive methotrexate IV over 24 hours on day 1, cytarabine BID IV over 3 hours on days 2 and 3, leucovorin IV or PO every 6 hours (Q6H) starting 12 hours after completion of methotrexate, filgrastim SC days 1-28, cytarabine IT on day 5-8 of cycles 2 and 4 and methotrexate IT on days 8-11 of cycles 2 and 4. Patients with CD20 expression may also receive rituximab IV on days 1 and 11 of cycles 1 and 3 and days 1 and 8 of cycles 2 and 4. Cycles repeat every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients may then receive DS-1594b PO BID on days 1-28, vincristine IV over 15 minutes on day 7 and prednisone PO BID on days 1-5. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 30 and 100.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written (signed) informed consent form (ICF) by the subject or legal guardian prior to the performance of any study-specific procedures, according to International Council on Harmonisation (ICH) and local regulatory requirements. Subject must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible toxicities) and must sign and date an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form (ICF)(including Health Insurance Portability and Accountability Act authorization [HIPAA], if applicable) before performance of any study-specific procedures or examinations
* Subjects must be willing and able to comply with the protocol
* Subjects with AML or ALL, diagnosed according to the 2016 criteria by the World Health Organization (WHO) who are refractory or relapsed (any salvage) with no available therapies or not candidates for available therapies. For subjects with prior MDS or chronic myelomonocytic leukemia (CMML) or MPN who transformed to AML, therapy received for MDS, CMML, or MPN is NOT considered as prior therapy for AML except for MDS or CMML treated with HMAs. Subjects with MDS or CMML treated with HMA therapies who progress to AML and have no available therapies or are not candidates for available therapies, will be eligible at the time of progression to AML. In Phase 1: all R/R AML or R/R ALL subjects irrespective of mutations will be eligible. In Phase 2 Cohort A only R/R AML with MLLr will be eligible. In Phase 2 Cohort B only R/R AML with NPM1m will be eligible. In Phase 2 Cohorts C and D: Only R/R AML or R/R ALL subjects with an MLLr or NPM1m will be eligible
* Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is permitted
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Total bilirubin =< 1.5 times upper limit of normal (x ULN)
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN (aspartate aminotransferase or alanine aminotransferase =< 5.0 x ULN if deemed related to leukemia by the treating physician)
* Creatinine clearance >= 50 mL/min as calculated using the modified Cockcroft-Gault equation
* Serum electrolytes within the institution's normal limits: potassium, calcium (total calcium, calcium corrected for serum albumin in case of hypoalbuminemia or ionized calcium) and magnesium. If outside of the institution's normal range, subject will be eligible when electrolytes are corrected
* In the absence of rapidly progressive disease, the interval from prior treatment to the time of initiation of protocol therapy will be at least 14 days for prior anti-leukemic therapy with the exception of hydroxyurea as noted below OR at least 5 half-lives for cytotoxic/noncytotoxic agents, whichever is shorter. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document. Since the effect of therapy may be delayed, use of hydroxyurea for subjects with rapidly proliferative disease is allowed before the start of study therapy and on study and hydroxyurea will not require a washout
* Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted. Subjects with a known history of CNS disease or leukemic brain metastasis must have been treated locally, have at least 3 consecutive lumbar punctures (LPs) with no evidence of CNS leukemia, and must be clinically stable for at least 4 weeks prior to enrollment and have no ongoing neurological symptoms that in the opinion of the treating physician are related to the CNS disease (sequelae that are a consequence of the treatment of the CNS disease are acceptable)
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 4 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
  * Combination of any of the two following (a+b or a+c or b+c)

    * a. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    * b. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * c. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
  * In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.
  * Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential

Exclusion Criteria:

* Subjects with a known allergy, hypersensitivity, or contraindication to the protocol therapies or any of their components to be used in the arm the subject is to be enrolled on
* Uncontrolled or significant cardiovascular disease, including any of the following:

  * Bradycardia of less than 50 beats per minute, unless the subject has a pacemaker;
  * Corrected QT interval Fridericia's Correction Formula (QTcF) interval > 450 msec;
  * Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
  * Systolic blood pressure >=180 mmHg or diastolic blood pressure >=110 mmHg;
  * History of clinically relevant ventricular arrhythmias within 6 months prior to screening (eg, ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes);
  * History of second (Mobitz II) or third-degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker);
  * History of uncontrolled angina pectoris, unstable angina or myocardial infarction, coronary artery bypass graft (CABG), cerebrovascular accident (CVA), transient ischemia attack (TIA), symptomatic pulmonary emboli within 6 months prior to screening;
  * New York Heart Association Class 3 or 4 heart failure;
  * Left ventricular ejection fraction (LVEF) =< 50 or less than the institutional lower limit of normal;
  * Complete left bundle branch block (right bundle branch block is permitted, but requires manual reading of the QTc interval);
  * Active cardiac dysrhythmias of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 (eg, atrial fibrillation)
* Persisting toxicity related to prior therapy of grade > 1 NCI-CTCAE v 5.0; however, alopecia and sensory neuropathy grade 2 or lower is acceptable
* Underwent HSCT within 90 days of the first dose of protocol therapy, or subjects with clinically significant (grade 2 or greater) graft-versus-host disease (GVHD) (the use of topical steroids for ongoing cutaneous GVHD is permitted)
* Subjects with symptomatic CNS leukemia or subjects with poorly controlled CNS leukemia
* Active and uncontrolled disease (active infection requiring systemic therapy, fever likely secondary to infection within prior 48 hours, uncontrolled hypertension despite adequate medical therapy as judged by the treating physician)
* Active (uncontrolled, metastatic) other malignancies
* Major surgery within 28 days prior to the first dose of protocol therapy
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (test at screening only if required by local regulations)
* Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with active Hepatitis B or C infection at screening (positive HBV surface antigen or HCV ribonucleic acid [RNA] if anti-HCV antibody screening test positive)
* Vaccination within 4 weeks of the first dose of study drug and while on trials is prohibited except for administration of inactivated vaccines
* Subjects who are currently receiving treatment with medication that meet one of the following criteria and that cannot be discontinued at least one week prior to the start of DS-1594b treatment:

  * Medications that may prolong QTc interval and have a known risk of inducing Torsades de Pointes unless it is vital for the care of the subjects
  * Strong inhibitors or inducers of CYP3A
  * CYP3A and CYP2C19 substrates with narrow therapeutic index
* Subjects who consume grapefruit products, Seville oranges, or star fruit within 3 days prior to the first DS-1594b administration and until the last day of DS-1594b is completed
* SUB-STUDIES: Subjects who are currently receiving moderate inhibitors or inducers of CYP3A who cannot discontinue at least one week prior to the start of DS-1594b treatment till the end of sub-study period
* SUB-STUDIES: Subjects who are currently receiving proton pump inhibitors who cannot discontinue at least 2 days prior to the start of DS-1594b treatment till the end of sub-study period
* Other severe acute or chronic medical conditions that is active and not well controlled including renal, skeletal muscle, adrenal insufficiency, colitis, inflammatory bowel disease, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Subjects unwilling or unable to comply with the protocol, including:

  * Pregnant or breastfeeding women or women of childbearing potential who are unable to comply with appropriate contraception as outlined in or who plan to become pregnant while in the study or for at least 6-7 months after last administration of study treatment
  * Known alcohol or drug abuse within the last 1 year
  * In a man whose sexual partner is a woman of childbearing potential, unwillingness or inability to use an acceptable contraceptive method for the entire study period and for at least 3 months after study completion
* Acute promyelocytic leukemia (APL)
* Uncontrolled or poorly controlled adrenal or pituitary disease (including adrenal insufficiency, Addison's disease, Cushing's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval G Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Numata M, Haginoya N, Shiroishi M, Hirata T, Sato-Otsubo A, Yoshikawa K, Takata Y, Nagase R, Kashimoto Y, Suzuki M, Schulte N, Polier G, Kurimoto A, Tomoe Y, Toyota A, Yoneyama T, Imai E, Watanabe K, Hamada T, Kanada R, Watanabe J, Kagoshima Y, Tokumaru E, Murata K, Baba T, Shinozaki T, Ohtsuka M, Goto K, Karibe T, Deguchi T, Gocho Y, Yoshida M, Tomizawa D, Kato M, Tsutsumi S, Kitagawa M, Abe Y. A novel Menin-MLL1 inhibitor, DS-1594a, prevents the progression of acute leukemia with rearranged MLL1 or mutated NPM1. Cancer Cell Int. 2023 Feb 25;23(1):36. doi: 10.1186/s12935-023-02877-y. PMID 36841758
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Groups:
- Phase I (DS-1594b) Cohort 1: Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  70 mg twice daily.
  DS-1594b: Given DS-1594b PO
- Phase I (DS-1594b) Cohort 2: Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  50 mg twice daily.
  DS-1594b: Given DS-1594b PO
- Phase I (DS-1594b) Cohort 3: Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  20 mg daily.
  DS-1594b: Given DS-1594b PO
- Phase I (DS-1594b) Cohort 4: Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  50 mg daily.
  DS-1594b: Given DS-1594b PO
- Phase I (DS-1594b) Cohort 5: Patients receive DS-1594b PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  100 mg daily.
  DS-1594b: Given DS-1594b PO
- Phase 2 Cohort A and B (DS-1594b): Patients with MLLr or NPM1m receive DS-1594b PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  DS-1594b: Given DS-1594b PO
- Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine): Patients receive DS-1594b PO BID on days 1-28, venetoclax PO QD on days 1-28, and azacitidine IV or SC on days 1-7. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  DS-1594b: Given DS-1594b PO
  Azacitidine: Given IV or SC
  Venetoclax: Given PO
- Phase 2 Cohort D (DS-1594b, Mini-HCVD): Patients receive DS-1594b PO BID on days 1-28. For additional information, see trial description.
  DS-1594b: Given DS-1594b PO
  Cyclophosphamide: Given IV
  Cytarabine: Given IT
  Dexamethasone: Given PO or IV
  Filgrastim: Given SC
  Leucovorin: Given IV or PO
  Mesna: Given IV
  Methotrexate: Given IT
  Prednisone: Given PO
  Rituximab: Given IV
  Vincristine: Given IV
Period: Overall Study
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Started | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Completed | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD) | Total
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 10
  >=65 years | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 0 |  |  |  | 5
  Male | 3 | 3 | 3 | 2 | 1 |  |  |  | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Asian | 0 | 0 | 1 | 0 | 0 |  |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 |  |  |  | 3
  White | 4 | 4 | 2 | 2 | 1 |  |  |  | 13
  More than one race | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 3 | 1 |  |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: The highest dose of DS-1594b treatment that does not cause unacceptable side effects.
Time Frame: Day 28
Population: as for baseline characteristics
Measure: Number; unit: Milligrams
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Milligrams | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. |  |  |

2. Primary Outcome: Recommended Phase 2 Dose (RP2D) (Phase I)
Description: This will be selected based upon the cumulative safety, efficacy and PK data at the end of the Phase 1 portion when the maximum tolerated dose is found. This will be One dose level below the RP2D of DS-1594b from Phase 1.
Time Frame: Day 28
Population: as for baseline characteristics
Measure: Number; unit: Milligrams
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Milligrams | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. | NA — The maximum tolerated dose in phase I was not reached. insufficient number of participants with events, study terminated early. |  |  |

3. Primary Outcome: Number of Participants With Complete Remission (CR) and Complete Remission With Partial Hematologic Recover (CRh)With DS-1594b Monotherapy in (Phase II, Cohort A)
Description: AML Participants: (CR) is No circulating blasts, Neutrophils > 1.0 x 10 ^ 9/L OR Platelet Count > 100 x 10 ^ 9/L, Bone marrow aspirate and biopsy <5% blasts, No Auer rods, No extramedullary leukemia. (CRh) is defined No circulating blasts, Neutrophils >/= 0.5 x 10 ^ 9/L, Platelet Count >/= 50 x 10 ^ 9/L, Bone marrow aspirate and biopsy <5% blasts, No Auer rods. ALL Participants: (CR) is No circulating lymphoblast or extramedullary disease, No lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement. Trilineage hematopoiesis (TLH) and <5% blasts, Neutrophil count > 1.0 x 10 ^ 9/L, platelet count > 100 x 10 ^ 9/L, No recurrence for 4 weeks. (CRh) No circulating lymphoblast or extramedullary disease, No lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement. Trilineage hematopoiesis (TLH) and <5% blasts, Neutrophil count >/= 0.5 x 10 ^ 9/L, >/= 50 x 10 ^ 9/L, No recurrence for 4 weeks.
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Achieved CR/CRh With DS-1594b Monotherapy in R/R AML With Nucleophosmin 1 Mutation (NPM1m) (Phase II, Cohort B)
Description: AML Participants: (CR) is No circulating blasts, Neutrophils > 1.0 x 10 ^ 9/L OR Platelet Count > 100 x 10 ^ 9/L, Bone marrow aspirate and biopsy <5% blasts, No Auer rods, No extramedullary leukemia. (CRh) is defined No circulating blasts, Neutrophils >/= 0.5 x 10 ^ 9/L, Platelet Count >/= 50 x 10 ^ 9/L, Bone marrow aspirate and biopsy <5% blasts, No Auer rods.
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Achieved CR+CRh With DS1594b in Combination With Azacitidine and Venetoclax in R/R MLLr or R/R NPM1m AML (Phase II, Cohort C)
Description: as for outcome 4
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Who Achieved CR+CRh With DS1594b in Combination With Mini-HCVD in R/R ALL With MLLr (Phase II, Cohort D)
Description: ALL Participants: (CR) is No circulating lymphoblast or extramedullary disease, No lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement. Trilineage hematopoiesis (TLH) and <5% blasts, Neutrophil count > 1.0 x 10 ^ 9/L, platelet count > 100 x 10 ^ 9/L, No recurrence for 4 weeks. (CRh) No circulating lymphoblast or extramedullary disease, No lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement. Trilineage hematopoiesis (TLH) and <5% blasts, Neutrophil count >/= 0.5 x 10 ^ 9/L, >/= 50 x 10 ^ 9/L, No recurrence for 4 weeks.
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: CR+ Complete Remission With Incomplete Hematologic Recovery (CRi) Rate of DS-1594b in Combination With Mini-HCVD in R/R ALL With MLLr (Phase II Cohort D)
Description: as for outcome 6
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Composite CR (CRc) Rate
Description: Defined as CR + complete remission with incomplete blood count recovery (CRi), morphologic leukemia free survival (MLFS), partial remission (PR), and overall response rate of subjects with R/R AML and R/R ALL treated on single-agent or combinations of DS-1594b.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

9. Secondary Outcome: Participants With Morphologic Leukemia-free State (MLFS)
Description: AML Participants: Bone marrow < 5% myeloblasts, no auer rods, no extramedullary leukemia, neutrophil or platelet recovery is not required.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 4 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

10. Secondary Outcome: Participants With a Partial Response (PR)
Description: Partial remission (PR), Neutrophil count: >1.0 x109/L, Platelet count >100 x109/L, ≥ 50 % reduction in bone marrow blast from pretreatment baseline, but still ≥ 5%.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

11. Secondary Outcome: Number of Participants With a Response
Description: Defined as CR + CRi + MLFS + PR. Complete remission (CR), Peripheral blood counts: No circulating blasts, Neutrophil count: >1.0 x109/L, Platelet count >100 x109/L, Bone marrow aspirate and biopsy: < 5% blasts, No Auer rods, No extramedullary leukemia. CRi is the same as CR except Neutrophil count: <1.0 x109/L, OR Platelet count: <100 x109/L. MLFS is Bone marrow < 5% myeloblasts, No Auer rods, No extramedullary leukemia, Neutrophil or platelet recovery is not required. PR is Neutrophil count: >1.0 x109/L, Platelet count >100 x109/L, >/= 50 % reduction in bone marrow blast from pretreatment baseline, but still >/= 5%
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

12. Secondary Outcome: Duration of Response
Description: Response date to loss of response or last follow up.
Time Frame: Up to 2 years
Population: There were zero responses, therefore duration of response was not calculated. Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Time to First Response and Time to Best Response
Description: First response date to best response date.
Time Frame: Up to 2 years
Population: There were zero responses, therefore time from response to best response was not calculated. Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Rate of Durable Transfusion Independence (TI)
Description: TI is defined as the absence of red blood cell and platelet transfusions for a consecutive 56-day period during continued treatment.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

15. Secondary Outcome: Event-free Survival
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Up to the date of failure or death from any cause, approximately 2 years, 7 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Months | 1.8 [0.5 to 3.3] | 0.7 [0.1 to 1.2] | 1.2 [0.6 to 3.0] | 2.6 [1.9 to 4.6] | 0.8 [0.8 to 0.8] |  |  |

16. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.From the date of the treatment start to the date of death or to the date of last follow-up if patients are alive at the time of data collection
Time Frame: Up to the date of death or last follow-up, approximately 2 years, 7 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Months | 4.3 [0.5 to 6.7] | 1.9 [0.1 to 4.0] | 2.3 [1.1 to 8.5] | 6.2 [5.5 to 6.9] | 7.2 [7.2 to 7.2] |  |  |

17. Secondary Outcome: Mortality Rate
Description: Number of deaths to occur within 4 weeks from start of therapy to 4 weeks into therapy.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 1 | 1 | 0 | 0 | 0 |  |  |

18. Secondary Outcome: Mortality Rate
Description: Number of deaths to occur within 8 weeks from start of therapy to 8 weeks into therapy.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 1 | 2 | 2 | 0 | 0 |  |  |

19. Secondary Outcome: Number of Subjects Able to Proceed to Hematopoietic Stem Cell Transplantation (HSCT) Without Additional AML Therapy
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 1 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 |  |  |

20. Secondary Outcome: Median Duration to HSCT From the Initiation of Single-agent or Combinations of DS-1594b in Subjects With RR AML and R/R ALL
Description: Calculated time to HSCR for participants who went on to HSCT.
Time Frame: Up to 2 years
Population: Zero Participants went on to HSCT, therefore the median duration to HSCT was not done. Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to the date of failure or death from any cause, approximately 3 years 7 months.
Description: Participant were only enrolled in the phase 1 portion of this study. The study was terminated early and did not move on to Phase 2.
Arm/Group | Phase I (DS-1594b) Cohort 1 | Phase I (DS-1594b) Cohort 2 | Phase I (DS-1594b) Cohort 3 | Phase I (DS-1594b) Cohort 4 | Phase I (DS-1594b) Cohort 5 | Phase 2 Cohort A and B (DS-1594b) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) | Phase 2 Cohort D (DS-1594b, Mini-HCVD)
All-Cause Mortality (participants affected / at risk) | 2/4 | 3/4 | 2/5 | 0/3 | 0/1 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 3/3 | 1/1 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 3/3 | 1/1 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (DS-1594b) Cohort 1 (N=4) | Phase I (DS-1594b) Cohort 2 (N=4) | Phase I (DS-1594b) Cohort 3 (N=5) | Phase I (DS-1594b) Cohort 4 (N=3) | Phase I (DS-1594b) Cohort 5 (N=1) | Phase 2 Cohort A and B (DS-1594b) (N=0) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) (N=0) | Phase 2 Cohort D (DS-1594b, Mini-HCVD) (N=0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 3 (6) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (DS-1594b) Cohort 1 (N=4) | Phase I (DS-1594b) Cohort 2 (N=4) | Phase I (DS-1594b) Cohort 3 (N=5) | Phase I (DS-1594b) Cohort 4 (N=3) | Phase I (DS-1594b) Cohort 5 (N=1) | Phase 2 Cohort A and B (DS-1594b) (N=0) | Phase 2 Cohort C (DS-1594b, Venetoclax, Azacitidine) (N=0) | Phase 2 Cohort D (DS-1594b, Mini-HCVD) (N=0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BUN increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (General disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (3) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (5) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (4) | 1 (1) | 2 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (5) | 4 (8) | 5 (12) | 3 (8) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04752163/Prot_SAP_000.pdf